CLINICAL TRIAL: NCT06780670
Title: PSMAcTION: A Phase II/III, Open-label, International, Multicenter, Randomized Study of AAA817 Versus Standard of Care in the Treatment of Adult Participants With PSMA Positive Metastatic Castration-resistant Prostate Cancer Who Progressed on or After [177Lu]Lu-PSMA Targeted Therapy
Brief Title: Open-label Study Comparing AAA817 Versus Standard of Care in the Treatment of Previously Treated PSMA-positive mCRPC Adults Who Have Disease Progressed on or After [177Lu]Lu-PSMA Targeted Therapy
Acronym: PSMAcTION
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA817A12201; 2024-512342-42-00 (Other: EU CTIS)
Record Dates: First submitted 2024-12-17; First posted 2025-01-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: post [177Lu]Lu-PSMA targeted therapy; PSMA-positive; mCRPC adults; Metastatic castration-resistant prostate cancer; AAA817; [225Ac]Ac-PSMA-617; PSMA-based targeted therapy; Standard of Care; SOC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — (225)Ac-PSMA-617

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase II: AAA817 Dose B (Experimental): AAA817 will be given for a number of cycles; a cycle = 8 weeks
  Interventions: Drug: AAA817
- Phase III: Investigator's choice of SoC (Active Comparator): Participants will be given Standard of Care (SOC) treatment per Investigator's choice.
  Interventions: Drug: Investigators choice of SoC
- Phase II: AAA817 Dose A (Experimental): AAA817 Dose A will be given for a number of cycles: a cycle = 8 weeks
  Interventions: Drug: AAA817
- Phase III: Recommended Phase 3 Dose of AAA817 (Experimental): Rp3D of AAA817 will be given for a number of cycles; a cycle = 8 weeks
  Interventions: Drug: AAA817

INTERVENTIONS:
Drug: Investigators choice of SoC — The control treatment in Phase III is investigator's choice of SoC
  Arms: Phase III: Investigator's choice of SoC
Drug: AAA817 — The investigational treatment is AAA817
  Other Names: [225Ac]Ac-PSMA-617)
  Arms: Phase II: AAA817 Dose A
Drug: AAA817 — The investigational treatment is AAA817
  Other Names: [225Ac]Ac-PSMA-617)
  Arms: Phase III: Recommended Phase 3 Dose of AAA817
Drug: AAA817 — Investigational treatment is the Dose B of AAA817
  Other Names: [225Ac]Ac-PSMA-617
  Arms: Phase II: AAA817 Dose B

SUMMARY:
This is a Phase II/III study. Patient population is adult participants with PSMA-positive mCRPC who had treatments with androgen receptor pathway inhibitor (ARPI) and taxane-based chemotherapy and progressed on or after [177Lu]Lu-PSMA targeted therapy.

Treatment of interest: the investigational treatment is AAA817 regardless of subsequent anti-neoplastic treatment. The control treatment is investigator's choice of Standard of Care, regardless of subsequent anti-neoplastic treatment

DETAILED DESCRIPTION:
Study CAAA817A12201 consists of 2 parts: a randomized, open-label, international, multicenter, phase II study (Phase II) to collect more information to support the proposed dose of AAA817 and a randomized, open-label, international, multicenter, 2- arm phase III study (Phase III) aimed to evaluate the efficacy and safety of proposed dose of AAA817 vs. investigator's choice of standard of care (SoC) in the treatment of adult participants with PSMA-positive metastatic castration-resistant prostate cancer (mCRPC) who had treatments with ARPI and taxane-based chemotherapy, and progressed on or after [177Lu]Lu-PSMA targeted therapy. The purpose of the phase II part (Phase II) of this study is to collect additional information to support proposed phase III dose of AAA817.

ELIGIBILITY:
Inclusion Criteria: ∙

* adults ≥ 18 years of age.
* ECOG performance status of 0 to 2.
* histopathological and/or cytological confirmation of adenocarcinoma of the prostate.
* PSMA-positive disease as assessed by PSMA PET/CT scan using an approved PSMA imaging agent as protocol instructed,
* castrate level of serum/plasma testosterone (< 50 ng/dL or < 1.7 nmol/L).
* Prior treatments with an androgen receptor pathway inhibitor (ARPI) and taxane-based chemotherapy, and progressed on or after [177Lu]Lu-PSMA targeted therapy.
* ≥ 1 metastatic lesion that is present on screening/baseline CT, MRI, or bone scan imaging obtained ≤ 28 days prior to randomization
* eGFR as requested by the sponsor

Exclusion Criteria:

* Any investigational agents within 28 days prior to the day of randomization.
* Any 225Ac-based investigational compound used prior to the day of randomization.
* Participants with a history of CNS metastases who are neurologically unstable, symptomatic, or receiving corticosteroids for the purpose of maintaining neurologic integrity.
* Concurrent acute kidney injury (renal failure developed between 48 hours to 7 days) or chronic kidney disease (at least 3 months of ongoing renal injury)
* Baseline xerostomia ≥ Grade 2 by CTCAE v.5
* History of uncontrolled hypertension, myocardial infarction (MI), angina pectoris, or coronary artery bypass graft (CABG) within 6 months prior to ICF signature and/or clinically active significant cardiac disease
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for basal cell carcinoma or actinic keratosis that have been treated with no evidence of recurrence in the past 3 months, non-invasive malignant colon polyps that have been removed).

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2028-06-27 (Estimated); Study Completion 2033-07-19 (Estimated)

PRIMARY OUTCOMES:
Biochemical response rate (Phase II) | from date of randomization up to approximately 24 months
  Biochemical response rate as defined as the percentage of participants who achieved a ≥ 50% decrease from baseline that is confirmed by a second measurement
Adverse Events (AEs) and Serious Adverse Events (SAEs), and deaths - Phase II | from day of randomization to 30 days after End of Treatment or (last AAA817 dose date + 55 days, last dose date of SoC + 30 days), whichever is later
  Safety defined as the type, incidence and severity of AEs and SAEs, and deaths
Tolerability of the proposed dose of AAA817- Phase II | From on-treatment period which start from the first dose of study treatment until 30 days post-last dose date for SoC and 55 days post last-dose for AAA817
  Percentage of participants who experienced Dose interruptions, reductions, discontinuation, dose intensity and duration of exposure
Radiographic progression-free survival (rPFS)- Phase III | from date of randomization up to approximately 24 months
  Percentage of participants who are alive without radiographic progression or who are lost to follow-up at the time of analysis
Overall survival (OS)- Phase III | from date of randomization up to approximately 24 months
  Percentage of participants who are alive or who are lost to follow-up at the time of analysis

SECONDARY OUTCOMES:
Radiographic progression-free survival (rPFS)- Phase II | from date of randomization up to approximately 24 months
  Percentage of participants who are alive without radiographic progression or who are lost to follow-up at the time of analysis
Progression free survival (PFS)- Phase II | from date of randomization up to approximately 24 months
  Percentage of Participants meeting Progression Free Survival
Overall response rate (ORR)- Phase II | from date of randomization up to approximately 24 months
  Percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR)
Disease control rate (DCR)- Phase II | from date of randomization up to approximately 24 months
  Percentage of participants with BOR of CR, PR, stable disease (SD) or non-CR/non-PD
Overall survival (OS)- Phase II | from date of randomization up to approximately 24 months
  Percentage of participants who are alive or who are lost to follow-up at the analysis data cut-off
Progression free survival (PFS) -Phase III | from date of randomization up to approximately 24 months
  Percentage of participants with PFS -defined as the time from date of randomization to first documented progression
Overall response rate (ORR)- Phase III | from date of randomization up to approximately 24 months
  ORR is defined as the percentage of participants with best overall response (BOR) of confirmed complete response (CR) or partial response (PR)
Disease control rate (DCR) -Phase III | from date of randomization up to approximately 24 months
  DCR is defined as the percentage of participants with BOR of confirmed CR, PR, stable disease (SD) or Non-CR/Non progressive disease (PD)
Duration of response (DoR)- Phase III | from date of randomization up to approximately 24 months
  Percentage of participants with confirmed DoR defined as duration of time between the date of first documented response (CR or PR) and progression or death due to any cause, whichever occurs first.
Time to first radiographic soft tissue progression (TTSTP)- Phase III | from date of randomization up to approximately 24 months
  Percentage of participants with confirmed first radiographic progression in soft tissue
First symptomatic skeletal event (TTSSE)_Phase III | from date of randomization up to approximately 24 months
  Percentage of participants with confirmed skeletal event is defined as new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, or requirement for radiation therapy to relieve bone pain, or death due to any cause, whichever occurs first
Prostate specific antigen (PSA) response -Phase III | from date of randomization up to approximately 24 months
  PSA50 is defined as the percentage of participants who achieved a confirmed ≥ 50% decrease from baseline
Patient reported disease related symptoms and health-related quality of life (HRQoL): Phase III | from date of randomization up to approximately 24 months
  Percentage of participants who had a Change from baseline on FACT-P Prostate Cancer Subscale (PCS)
Time to worsening on the Worst Pain: Phase III | from date of randomization up to approximately 24 months
  Time to worsening on the Worst Pain defined as the time from randomization to the first occurrence of worsening on the Worst Pain item (brief pain inventory - short form (BPI-SF)) of at least 30% of baseline or minimum of 2 points increase from baseline, or death due to any cause, whichever occurs first. BPI-SF is a self-reported questionnaire to evaluate pain intensity (severity) and impact of pain on the participant's daily functioning (interference).

CONTACTS AND LOCATIONS:
Locations (27):
- United States (3):
  - Indiana University, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - WA Uni School Of Med, St Louis, Missouri
- Australia (2):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Herston, Queensland
- Novartis Investigative Site, São Paulo, São Paulo, Brazil
- China (6):
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Japan (7):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Kyoto
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Novartis Investigative Site, Taipei, Taiwan